CLINICAL TRIAL: NCT05900973
Title: A Phase 2 Trial of Darolutamide as a Prostate-Specific Membrane Antigen (PSMA) Expression Enhancer in Patients With Localized Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: D'Or Institute for Research and Education (Other)
Collaborators: Bayer (Industry); RPH Central Pharma (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ID 389-22-ONCO-FOMENTO-SP
Record Dates: First submitted 2023-05-08; First posted 2023-06-13 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; PET PSMA; Prostate-specific membrane antigen (PSMA); Darolutamide
MeSH Terms: conditions — Prostatic Neoplasms | interventions — darolutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NUBEQA® (darolutamide) administered to participants (Experimental): Oral use of Darolutamide as an Inducer of Increased Expression of Prostate-specific membrane antigen (PSMA) in patients with Localized prostate cancer
  Interventions: Drug: Darolutamide Oral Tablet [Nubeqa]

INTERVENTIONS:
Drug: Darolutamide Oral Tablet [Nubeqa] — Oral use of Darolutamide as an Inducer of Increased Expression of Prostate-specific membrane antigen (PSMA) in patients with Localized prostate cancer

SUMMARY:
Prostate cancer is the second leading cause of cancer death in men. According to estimates by the American Cancer Society Prostate for 2022, about 268,490 men would be diagnosed with prostate cancer and 34,500 would die from the disease. Clinical evolution follows the clinical stages are: localized disease, biochemical recurrence after surgery or radiotherapy, and castration-sensitive or castration-resistant metastatic disease. Localized disease is often classified according to a risk stratification system, which includes assessment of the Gleason score, prostate-specific antigen (PSA) at diagnosis, number of involved fragments per disease at biopsy, and clinical T-staging. Gleason score greater than or equal to 8, PSA greater than or equal to 20 ng/dL at diagnosis, and/or involvement of the prostatic capsule or seminal vesicle are high-risk criteria for biochemical recurrence and later development of metastases, for which the standard treatment is radical prostatectomy or radiotherapy plus androgen deprivation therapy. Prostate-specific membrane antigen (PSMA) is highly expressed on the surface of prostate cancer cells, with relatively low expression in normal tissue. PSMA has been explored as a target in imaging studies using positron emission tomography (PSMA-PET) to reveal occult metastatic disease, as well as a target in the development of PSMA-based treatments with radioligands. According to Hoffman et al., performing PSMA-PET demonstrated greater sensitivity (85% vs. 38%) and specificity (98% vs. 91%), and determined more changes in patient management (28% vs. 15% ) compared to conventional images. Other studies have also demonstrated the greater accuracy of PSMA-based radiotracers compared to conventional images. Finding strategies that increase PSMA expression is a necessity for patients with prostate cancer. According to researchers, high SUVmax values are associated with better outcomes in patients treated with 177-lutetium-PSMA-617. PSMA expression can be rapidly modulated by androgen suppression. The investigators understand that there is great potential to evaluate darolutamide as a PSMA expression enhancer. However, to date there are no prospective data evaluating the effect of ARSI in increasing PSMA expression in localized disease. Here the investigators propose a phase 2 study to investigate the efficacy of a limited course of darolutamide as a PSMA expression enhancer in men with localized prostate cancer according to conventional imaging. PSMA-PET/CT scans will be acquired before and after treatment with darolutamide, as detailed in the protocol. Slides of prostate biopsies and prostatectomies stained with hematoxylin and eosin (H&E) will be reviewed by two pathologists to select the most representative tumor block. Immunohistochemical (IHC) reaction using standard protocols will be performed using an anti-PSMA antibody and intraprostatic anti-androgens. Gene expression analysis will be performed using RNA extracted from biopsies and prostatectomies and evaluated by a panel of over 300 transcripts. For methylation patterns, hematoxylin and eosin (H&E) slides from prostate biopsies and prostatectomies will undergo DNA extraction and evaluation of the methylation profile performed using a kit. It is expected to identify that treatment with darolutamide increases PSMA expression and that the biochemical mechanisms involved can be better evidenced.

ELIGIBILITY:
Inclusion Criteria

* To be included in this study, patients should complete all screening procedures and meet all of the following criteria:
* Males 18 years of age and above
* Histologically or cytologically proven diagnosis of prostate adenocarcinoma
* High-risk disease defined as at least one of the following factors:
* Gleason ≥8
* PSA ≥20 ng/mL
* T3/T4 disease
* ECOG Performance status of 0 or 1 (Appendix A: Performance Status Criteria)
* Patients deemed appropriate candidates for radical prostatectomy
* Baseline blood pressure <160 x 100 mmHg
* Normal hematologic, liver, and renal functions
* Absence of any contraindications for darolutamide use
* Willing and able to provide, or have a legally authorized representative provide, written informed consent and HIPAA authorization for the release of personal health information. A signed informed consent must be obtained before screening procedures are performed.
* Baseline testosterone of 200 ng/dL or more
* Normal organ function with acceptable initial laboratory values within 14 days of treatment start: Match lab values to those scheduled in Table 1.
* ANC • > 1,500/µl
* Hemoglobin • > 9g/dL
* Platelet count • > 100,000/µl
* Creatinine • ≤ 1.5 x the institutional upper limit of normal (ULN)
* Potassium • > 3.5 mmol/L (within institutional normal range)
* Bilirubin • ≤ ULN (unless documented Gilbert's disease)
* SGOT (AST) • ≤ 2.5 x ULN
* SGPT (ALT) • ≤ 2.5 x ULN

Exclusion Criteria

* Metastatic disease defined by standard scans (bone scans, magnetic resonance, or CT scans)
* Any prior or current treatment for prostate cancer
* Concomitant treatment with another systemic antineoplastic therapy or another investigational product is prohibited, as follows:
* Any investigational product
* Radiopharmaceuticals
* Immunotherapy (e.g. sipuleucel-T)
* Prior orchiectomy or any LHRH agonist or antagonist
* Cytotoxic chemotherapy
* Enzalutamide, apalutamide, bicalutamide, flutamide, nilutamide
* Estrogens
* Cyproterone acetate
* 5-alpha-reductase inhibitors
* Abiraterone acetate, TAK-700 or other CYP17 inhibitors
* Systemic ketoconazole
* Any drug listed in Appendix C
* Patients on current treatment for a second malignancy (except for Ta bladder urothelial carcinoma or non-melanoma skin cancer).
* Uncontrolled hypertension (defined as systolic blood pressure of 150 mmHg or higher; diastolic blood pressure of 100 mmHg or higher in 2 or more measurements) or uncompensated cardiac disease (NYHA III or IV)
* Known allergy, hypersensitivity, any other contraindications to the compounds under investigation (darolutamide or PSMA radiotracers)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males 18 years of age and above, histologically or cytologically proven diagnosis of prostate adenocarcinoma
Enrollment: 19 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2025-05-17 (Estimated); Study Completion 2025-05-24 (Estimated)

PRIMARY OUTCOMES:
Intraindividual pre- and post-treatment SUVmax. | 7 days
  The proportion of patients achieving an increase in the SUVmax of 20% or higher will be reported with two-sided 90% confidence interval (corresponding to the one-sided α=0.05 in the statistical design) that accounts for the two-stage design.

SECONDARY OUTCOMES:
Increase of PSMA-PET/CT parameters | 7 days
  PSMA PET/CT pre- and post-treatment will also be reported with 90% exact binomial CI.
Detection rate of extrapelvic metastatic disease pre- and post-darolutamide | 7 days
  The proportion of patients with planned management changes accordingly to PSMA PET/CT pre- and post-treatment will also be reported with 90% exact binomial CI. Any lesion with an SUV greater than the hepatic background will be considered a PSMA-positive lesion.
Detection rate of pelvic nodal metastatic disease pre- and post- darolutamide. | 7 days
  The proportion of patients with planned management changes accordingly to PSMA PET/CT pre- and post-treatment will also be reported with 90% exact binomial CI. Any lesion with an SUV greater than the hepatic background will be considered a PSMA-positive lesion.
Proportion of planned management changes with PSMA PET pre- and post- darolutamide. | 7 days
  The proportion of patients with planned management changes accordingly to PSMA PET/CT pre- and post-treatment will also be reported with 90% exact binomial CI. Treatment decisions will be made at physician's discretion.

OTHER OUTCOMES:
Immunochemical expression of PSMA and to correlate with PSMA-PET/CT parameters. | 7 days
  Findings in immunohistochemistry in PSMA will be reported using descriptive statistics. Pre- and post-treatment IHC measures will be summarized according to results of biopsy and prostatectomy pathology, whenever available.
To evaluate the pre- and post-treatment levels of intraprostatic androgens and to correlate with PSMA-PET/CT parameters. | 7 days
  PSA and testosterone levels:
  Findings in PSA and testosterone levels will be reported using descriptive statistics. Pre- and post-treatment measures will be summarized according to results of biopsy and prostatectomy pathology, whenever available.
  Intraprostatic androgens:
  Findings in intraprostatic androgen levels will be reported using descriptive statistics. Pre- and post-treatment measures will be summarized according to results of biopsy and prostatectomy pathology, whenever available.
To evaluate the pre- and post-treatment methylome patterns and to correlate with PSMA-PET/CT parameters. | 7 days
  Findings in immunohistochemistry in PSMA will be reported using descriptive statistics. Pre- and post-treatment IHC measures will be summarized according to results of biopsy and prostatectomy pathology, whenever available.

CONTACTS AND LOCATIONS:
Overall Officials: José Mauricio SC Mota, phD, Principal Investigator — Instituto D'Or de Pesquisa e Ensino (IDOR), São Paulo, Brazil
Locations (1):
- Instituto D'Or de Pesquisa e Ensino, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Records must be retained and securely stored until: (a) two (2) years after the date of approval of a new drug application for the study drug that is the subject of the clinical trial; or (b) two (2) years after the investigational new drug order for such study drug is closed or withdrawn, or for such longer period of time as may be required by participant policies, applicable laws, rules or regulations.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 05/20/2023 - 05/26/2027
Access Criteria: The data obtained by the study will be shared by the IT sector electronically by allowing researchers to access file folders stored on the host institution's server.
  There are no restrictions on sharing the data included in the study between the researchers involved.